CLINICAL TRIAL: NCT00419861
Title: Inpatient Surveillance for Influenza Infections in Adults
Brief Title: Inpatient Influenza Surveillance
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0051
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: Influenza, surveillance, flu, parent protocol
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal and throat swabs will be obtained and combined for viral culture, rapid antigen testing, and PCR. Specimens obtained from hospitalized subjects will be tested for influenza A & B viruses by viral culture, rapid antigen testing and Real-Time Reverse-Transcriptase PCR (RTrtPCR) analysis.

GROUPS / COHORTS (1):
- Group 1: Adults >/= 50 years of age, hospitalized for respiratory illness in Davidson County, TN.

SUMMARY:
Influenza vaccination is recommended for all persons age 65 and older. Vaccines that are designed and tested in young healthy adults are often not as effective when used in the elderly. This study will be a one year pilot study to see if it would be practical to conduct a larger study at several other hospitals in the future. Study participants will include 350 men and women greater than or equal to age 50 that are hospitalized at Vanderbilt University or Baptist Community Hospital with acute respiratory symptoms. Study procedures will include questions, one nasal swab, one throat swab, and chart reviews after the patient has been released from the hospital. The nasal and throat swabs will be tested for influenza A and B viruses.

DETAILED DESCRIPTION:
Influenza vaccination has been recommended for all persons greater than or equal to age 65, recent studies have questioned the efficacy of the vaccine in the aging population. The willingness to test new vaccines depends on a convincing demonstration of a significant burden of disease despite current vaccine policies. If comprehensive surveillance could be performed in a well defined population of adults over 50 years of age hospitalized with acute respiratory illness or fever, the precise burden of influenza illness in this age group could be determined and the risk factors associated with influenza infection established. This study will be a one year pilot study. Study participants will include 350 adults greater than and equal to 50 years of age hospitalized at Vanderbilt University or a local community hospital, Baptist Hospital, with acute respiratory symptoms or fever. The purpose of the study is to determine the feasibility of conducting a larger surveillance study in several other hospitals. Specific aims are: 1) to perform population-based surveillance to determine the etiology and burden of acute viral respiratory diseases or fever among hospitalized adults greater than or equal to 50 years of age and 2) to identify risk factors associated with hospitalization for vaccine-preventable respiratory disease in adults greater than or equal to 50 years of age. During November 2006 through April 2007, recruitment will occur 2 days per week and will increase to 4 days per week during the defined influenza season based on local surveillance. Following informed consent, there will be 3 parts to data collection: (1) series of brief questions; (2) one nasal and one throat swab will be collected and; (3) chart abstractions performed after discharge. Nasal and throat swabs will be tested for influenza A and B viruses by both viral culture, rapid antigen testing, and Real-Time Reverse-Transcriptase PCR (RTrtPCR) analysis. The primary endpoint of the study is the incidence of hospitalizations due to influenza virus by age, sex, and race in adults greater or equal to than 50 years of age. This study is linked to DMID protocol 06-0092.

ELIGIBILITY:
Inclusion Criteria:

1. Adults greater than or equal to 50 years of age
2. Resident of Davidson County
3. Admitted to hospital during defined 24 hour periods
4. Patients with one or more of the following admission diagnoses: pneumonia, upper respiratory infection, bronchitis, influenza, chronic obstructive pulmonary disease, asthma, viral illness, dyspnea, acute respiratory failure, pneumonitis due to solids/liquids, or fever without localizing symptoms

Exclusion Criteria:

1. Adults greater than or equal to 50 years residing outside the surveillance areas
2. Adults greater than or equal to 50 years not admitted on a surveillance day
3. Adults < 50 years of age

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  1. Adults >/= 50 years of age
  2. Resident of Davidson County
  3. Admitted to hospital during defined 24 hour periods
  4. Patients with one or more of the following admission diagnoses (International Classification of Diseases, 9th Revision Number): pneumonia (480-486), upper respiratory infection (465), bronchitis (466), influenza (487), chronic obstructive pulmonary disease (490 to 492;496), asthma (493), viral illness (079.9)[13], dyspnea (786), acute respiratory failure (518.81), pneumonitis due to solids/liquids (507), or fever (780.6) without localizing symptoms.
  Exclusion Criteria:
  1. Adults >/= 50 years residing outside the surveillance areas
  2. Adults >/= 50 years not admitted on a surveillance day
  3. Adults < 50 years of age
  4. Anyone without the above admitting criteria.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States